CLINICAL TRIAL: NCT01329016
Title: Glyburide and Metformin for Gestational Diabetes Mellitus
Brief Title: Glyburide and Metformin for Gestational Diabetes Mellitus (GDM)
Acronym: GDM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Washington (Other); University of Pittsburgh (Other); University of Texas (Other); Indiana University School of Medicine (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 820
Record Dates: First submitted 2011-03-22; First posted 2011-04-05 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Pregnancy; Glyburide; Metformin; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glyburide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GDM Subjects (Active Comparator): Women with GDM requiring treatment
  Interventions: Drug: Glyburide; Drug: Metformin; Drug: Glyburide-Metformin combination
- Non-pregnant Type 2 Diabetes Milletus Subjects (No Intervention): Non-pregnant women with Type 2 diabetes mellitus who plan to use metformin treatment
- Healthy Pregnant Women (No Intervention): Healthy pregnant women with normal 1-hour glucose tolerance test

INTERVENTIONS:
Drug: Glyburide — Women with GDM who require treatment will be given glyburide 2.5 mg. Medication will be given at least twice daily and equal doses will be given for each dosing time for the 3 days prior to the pharmacokinetic study day.
  Arms: GDM Subjects
Drug: Metformin — Women with GDM requiring treatment will be given metformin 500 mg. Medication will be administered at least twice daily and equal doses will be given for each dosing time for the 3 days prior to the pharmacokinetic study day.
  Arms: GDM Subjects
Drug: Glyburide-Metformin combination — Women with GDM requiring treatment will be given glyburide 2.5 mg with metformin 500 mg. Medications will be administered at least twice daily and equal doses will be given for each dosing time 3 days prior to the pharmacokinetic study day.
  Arms: GDM Subjects

SUMMARY:
This is a pharmacokinetic and pharmacodynamic study evaluating glyburide, metformin, and combination treatment for gestational diabetes mellitus.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is a common complication of pregnancy. Multiple treatment regimens are currently used for the management of GDM. Following failure of diet therapy, insulin, glyburide and metformin are all used in the treatment of GDM with the oral medications providing comparable outcomes with insulin but easier route of administration and schedule. The proposed work will evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of glyburide and metformin alone and in combination in order to lay the foundation in establishing dosage and response information that could be utilized in designing a phase III randomized trial that will ultimately evaluate GDM treatment optimization.

ELIGIBILITY:
Inclusion Criteria:

Gestational Diabetes Subject Selection

1. Pregnant women (singleton pregnancy)
2. Gestational diabetes mellitus
3. Able to give written informed consent
4. Drug treatment is required for GDM
5. Gestational age 20-32 weeks

   * Gestational diabetes diagnosis must occur after 20 weeks and prior to 32 weeks gestation
   * Randomization and treatment initiation must occur no later than 32 weeks gestation
6. Willing to avoid ethanol
7. 18-45 years of age

Type 2 Diabetes Mellitus Subject Selection

1. Able to give written informed consent
2. New diagnosis of type 2 diabetes mellitus
3. Plan to receive metformin for treatment of type 2 diabetes mellitus
4. 18-45 years of age
5. Female
6. Negative pregnancy test
7. Hemoglobin A1C > 7%

Healthy Pregnant Women

1. Able to give written informed consent
2. Pregnant women (singleton)
3. Normal 1-hour glucose tolerance test
4. 20-32 weeks gestation
5. 18-45 years of age

Neonates: All the infants of the pregnant women participating in this study will be included

Exclusion Criteria:

Women with GDM and T2DM

1. Women taking medications expected to interact with glyburide, metformin or alter blood glucose concentrations
2. Serum creatinine > 1.2 mg/dL
3. Hematocrit < 28%
4. Allergy to glyburide, metformin or sulfa
5. Significant hepatic disease
6. Congestive heart failure or history of MI
7. Moderate to severe pulmonary disease
8. Adrenal or pituitary insufficiency

Healthy Pregnant Women

1. Receiving any hypoglycemic agents
2. Receiving corticosteroids
3. Known kidney, liver, heart, pulmonary, adrenal or pituitary disease
4. Hematocrit < 28%

Neonates

1. Infants that are not viable or too ill for blood sample collection will be included for clinical outcomes data collection, but will be excluded from other research activities.
2. Infants < 1.5 kg will be included for clinical outcomes data collection, but will be excluded from blood sample collection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Study drug dosage in pregnancy | Completion of data collection (4-5mnths on average in GDM and healthy pregnant women and max of 6 months in newly diagnosed T2DMs)
  (1) Determination of metformin dosage in pregnancy needed to produce comparable concentrations to the approved dosage range in non-pregnant women. (2)To compare metformin apparent oral clearance in pregnant and non-pregnant women. (3)To evaluate the effect of GLY monotherapy, MET monotherapy, and GLY-MET combination on insulin sensitivity, beta-cell responsivity index and disposition index (response vectors) describing the mechanism and magnitude of effect.

SECONDARY OUTCOMES:
Determine GLY and MET PK parameters | Conclusion of data collection (up to 6 months)
  Determining GLY & MET PK parameters, including AUC, max concentration, time to max & min concentrations, oral clearance, half-life, oral volume of distribution, umbilical cord plasma concentrations; correlation between CYP2C9, CYP3A5, BCRP, OATP2B1 genotypes & GLY PK/PD; GLY & MET PD parameters, including derived parameters from PK/PD modeling for pregnant & nonpregnant subjects; duration of initiation of treatment to glycemic control; effects of GDM & glycemic control on maternal & umbilical cord EPC cells & sFLT concentrations; GLY & MET half-life in neonates; efficacy & safety data.

CONTACTS AND LOCATIONS:
Overall Officials: Mary F. Hebert, PharmD, FCCP, Principal Investigator — University of Washington; Steve Caritis, MD, Principal Investigator — University of Pittsburgh; Gary DV Hankins, MD, Principal Investigator — University of Texas; David Flockhart, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington, Seattle, Washington